CLINICAL TRIAL: NCT00570115
Title: Left Atrial Volume and Function in Patients With Obstructive Sleep Apnea Assessed by Real Time Three Dimensional Echocardiography
Brief Title: Left Atrial Volume and Function Evaluation in Patients With Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Wercules Antonio Alves de Oliveira, AFIP/Instituto do Sono
Other Study IDs: ecoera-001
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2007-12

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sleep Apnea Syndromes diastolic disfunction left atrium
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: The subjects for this group are matched for age, gender, body mass index. The presence of obstructive sleep apnea will divide the cohort in 02 subgroups: non-Obstructive Sleep Apnea and Obstructive Sleep Apnea

SUMMARY:
The purpose of this study is to determine whether patients with obstructive sleep apnea have any changes in left atrial morphology and function evaluated by echocardiography three dimensional

DETAILED DESCRIPTION:
Several studies have been suggesting that Obstructive Sleep Apnea contributes to deterioration of left ventricular diastolic function . It may lead to atrial myocardium stretching and enlargement which may be associated to increased risk of cardiovascular events. We hypothesized that morphological and functional LA changes might be found using three dimensional echo, and that such alterations are related to obstructive sleep apnea presence.

ELIGIBILITY:
Inclusion Criteria:

* Age from 30 to 70
* Apnea-hypopnea index > 5 by polysomnography

Exclusion Criteria:

* Any cardiac disease
* Poor imaging quality by mean of echocardiography
* non-sinusal Rhythm

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators recruited 56 recently diagnosed OSA patients, confirmed by full polysomnography (PSG), referred to Sleep Laboratory of Psychobiology Department of Federal University of Sao Paulo, Brazil, according to the following inclusion criteria: both genders aging from 29 to 70 years old, with apnea-hypopnea index (AHI) >5 events/hour of sleep. Control group comprised 50 healthy community subjects without OSA confirmed by full PSG, matched by age, gender, and BMI.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2007-06; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Left Atrial enlargement | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Tufik, PhD,MD., Study Director — Federal University of São Paulo
Locations (1):
- Instituto do Sono/Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Anwar AM, Soliman OI, Geleijnse ML, Nemes A, Vletter WB, ten Cate FJ. Assessment of left atrial volume and function by real-time three-dimensional echocardiography. Int J Cardiol. 2008 Jan 11;123(2):155-61. doi: 10.1016/j.ijcard.2006.12.017. Epub 2007 Apr 17. PMID 17442422